CLINICAL TRIAL: NCT03722121
Title: Is the Distance of Patients From Rouen University Hospital Influencing the Time Between Colectomy and First Chemotherapy Cure for Colon Cancer?
Acronym: DICHIMIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/264/HP
Record Dates: First submitted 2017-10-27; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Cancer Colon; Colectomy; Chemotherapy
Keywords: distance
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project has for objective to demonstrate that the increase of the distance "Patient home - center of treatment" may be associated with significant, other noticeable, noted events. This distance may also be available in the Rouen University Hospital. The study of the association in this distance and the delay in initiating chemotherapy after surgery in patients treated at the CHU correspond to a pilot study prior to the completion of the analysis at the regional scale.

ELIGIBILITY:
Inclusion Criteria:

- Patients who had colectomy for colon cancer and at least one chemotherapy treatment at CHU Rouen, between 2009 and the first half of 2015.

Exclusion Criteria:

* Patients who died in hospital before receiving a chemotherapy treatment
* Patients with a CIM code of metastasis during the stay of the colectomy or the first chemotherapy treatment
* Patients who received a chemotherapy treatment before colectomy
* Patients who have undergone several colectomies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient having a cancer colon and hospitalized for colectomy: malignant tumor colon, in situ colon carcinoma or tumor with unpredictable or unknown evolution of the colon
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-12-23 (Estimated)

PRIMARY OUTCOMES:
distance "home of patients - treatment center" | At the inclusion
  Analyze the influence of distance "home of patients - treatment center" on the compliance of the time between colectomy and initiation of CTa

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France